CLINICAL TRIAL: NCT01023685
Title: An Open-label Extension to a 52-week, Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel Group Study in Patients With Alzheimer's Disease to Investigate the Safety and Tolerability of Repeated Subcutaneous Injections of CAD106.
Brief Title: To Investigate the Safety and Tolerability of Repeated Subcutaneous Injections of CAD106 in Alzheimer's Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCAD106A2202E1
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2013-06

CONDITIONS: Alzheimer Disease
Keywords: Active immunization; Alzheimer disease; Antibody; Central Nervous System diseases; Neurodegenerative diseases; Vaccine
MeSH Terms: conditions — Alzheimer Disease; Central Nervous System Diseases; Neurodegenerative Diseases

ARMS (1):
- CAD106 (Experimental)
  Interventions: Biological: CAD106

INTERVENTIONS:
Biological: CAD106

SUMMARY:
This study will investigate the Safety and Tolerability of Repeated Subcutaneous Injections of CAD106 in Alzheimer's Patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed the core study with no significant safety concerns

Exclusion Criteria:

* Diagnosis of other neurodegenerative disease and/or psychiatric disorders (with the exception of successfully treated depression).
* Diagnosis or presence of an active, uncontrolled seizure disorder and/or cerebrovascular disease.
* Diagnosis or presence of an active autoimmune and/or with an acute or chronic inflammation.

Other protocol-defined inclusion/exclusion criteria may apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Safety/tolerability assessments at multiple time points including but not limited to screening, and through to the end of the study to week 66. | 66 weeks

SECONDARY OUTCOMES:
Collect long-term safety information through SAE's collection for two years after completion of the extension study. | 2 years
Immune response, cognitive and functional assessments at multiple time points including but not limited to baseline, and through to the end of the study to week 66. | 66 weeks
Evaluate the antibody response after 4 additional injections in the Extension study, in patients initially treated with CAD106 in the Core study. | 66 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- United States (8):
  - ATP Clinical Research, Inc., Costa Mesa, California
  - Alpin Research Center, Boulder, Colorado
  - Sunrise Clinical Research, Inc., Hollywood, Florida
  - Alexian Brothers Neuroscience Institute, Elk Grove Village, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Volunteer Research Group, Knoxville, Tennessee
  - University of Texas Southwestern, Dallas, Texas

REFERENCES:
- [Derived] Farlow MR, Andreasen N, Riviere ME, Vostiar I, Vitaliti A, Sovago J, Caputo A, Winblad B, Graf A. Long-term treatment with active Abeta immunotherapy with CAD106 in mild Alzheimer's disease. Alzheimers Res Ther. 2015 Apr 27;7(1):23. doi: 10.1186/s13195-015-0108-3. eCollection 2015. PMID 25918556
- See also: Results for CCAD106A2202E1 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=8123